CLINICAL TRIAL: NCT02658318
Title: Postoperative Complications After Cleft Palate Closure in Patients With Pierre Robin Sequence: Operative Considerations
Status: Completed | Type: Observational
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Johan Abeloos, Maxillofacial surgeon, Head of Department, AZ Sint-Jan AV
Other Study IDs: B049201525560
Record Dates: First submitted 2016-01-11; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Pierre Robin Syndrome; Cleft Palate
Keywords: peri- and postoperative complications; airway obstruction; adapted Furlow palatoplasty
MeSH Terms: conditions — Pierre Robin Syndrome; Cleft Palate; Postoperative Complications; Airway Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pierre Robin Syndrome (PRS): Cleft palate patients with the Pierre Robin Syndrome.
- non-PRS: Cleft palate patients without the Pierre Robin Syndrome.

SUMMARY:
In cleft surgery there is no current general agreement on the treatment strategy of patients with the Pierre Robin Sequence. The timing of surgery and the surgical approach depends on the treating physician or the hospital facility. Literature regarding peri- and postoperative complications in the target population are lacking.

The investigators aim to retrospectively review the charts of all cleft patients, both PRS and non-PRS, treated with an adapted Furlow palatoplasty between 01/01/2011 and 31/08/2015. The incidence of peri- and postoperative complications, with a specific focus on respiratory complications, will be examined. The value of demographic, surgical and postoperative parameters will be examined as potential risk factors for the development of complications.

ELIGIBILITY:
Inclusion Criteria:

* patients of all ages
* patients that had undergone a modified Furlow palatoplasty
* patients treated at the GH Saint-John Bruges (Belgium), or the cooperating Semmelweis University (Hungary)

Exclusion Criteria:

* patients not eligible according to the abovementioned criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cleft patients consecutively treated with a modified Furlow palatoplasty between 01/01/2011 and 31/08/2015 in the Department of Oral and Maxillofacial Surgery of the General Hospital Saint-John Bruges (Bruges, Belgium) or the Department of Pediatrics of the Semmelweis University (Budapest, Hungary)
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2011-01; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Incidence of peri- and postoperative complications | within 4 weeks postoperative

SECONDARY OUTCOMES:
Identification of potential risk factors (demographic, diagnostic, surgical) for development of postoperative complications, through regression analysis | within 4 weeks postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Johan Abeloos, MD, Principal Investigator — Maxillofacial surgeon, Head of Department
Locations (1):
- General Hospital Saint-John Bruges, Bruges, Belgium

IPD SHARING:
Plan to Share IPD: No